CLINICAL TRIAL: NCT01775189
Title: A Randomized, Double-blind, Placebo Controlled, Single-dose, 4-way Crossover Study To Determine The Relative Abuse Potential Of Alo-02 (Oxycodone Hydrochloride And Naltrexone Hydrochloride Extended Release Capsules) Compared To Oxycodone Immediate Release, And Placebo When Administered Intranasally To Non-dependent, Recreational Opioid Users.
Brief Title: A Study to Characterize the Abuse Liability of ALO-02 in Healthy, Non-Dependent, Recreational Opioid Users When ALO-02 Capsules Are Crushed and Snorted
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: B4531009
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: Relative abuse potential study; Chronic pain; oxycodone; naltrexone; opioid-related disorders; drug abusers
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Drug Misuse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Placebo Comparator)
  Interventions: Drug: ALO-02 weight-matched placebo
- Treatment B (Experimental)
  Interventions: Drug: crushed ALO-02 30 mg/3.6 mg
- Treatment C (Placebo Comparator)
  Interventions: Drug: oxycodone weight-matched placebo
- Treatment D (Active Comparator)
  Interventions: Drug: crushed oxycodone IR 30 mg

INTERVENTIONS:
Drug: ALO-02 weight-matched placebo — crushed sugar spheres (powder) x 1 dose
  Arms: Treatment A
Drug: crushed ALO-02 30 mg/3.6 mg — crushed ALO-02 30 mg/3.6 mg capsule x 1 dose
  Arms: Treatment B
Drug: oxycodone weight-matched placebo — crushed lactose tablets (powder) x 1 dose
  Arms: Treatment C
Drug: crushed oxycodone IR 30 mg — Three (3) crushed immediate-release (IR) oxycodone 10 mg tablets x 1 dose
  Arms: Treatment D

SUMMARY:
The main purpose of this study is to determine if oxycodone and naltrexone combination capsules (ALO-02) have the potential to be abused when they are crushed and snorted.

DETAILED DESCRIPTION:
Abuse Liability Study

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Non-dependent, recreational opioid users. (Must use opioid for non-therapeutic purposes on at least 10 occassions within the last year and at least once in the 8 weeks before Visit 1 (Screening Visit).
* Must have experience with intranasal opioid administration (snorted opioid drugs on at least 3 occassions within the last year before Visit 1 (Screening Visit).

Exclusion Criteria:

* Diagnosis of substance and/or alcohol dependence
* Subject has participated in, is currently participating in, or seeking treatment for substance and/or alcohol related disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- INC Research Toronto Inc., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Setnik B, Bramson C, Bass A, Levy-Cooperman N, Malhotra B, Matschke K, Sommerville KW, Wolfram G, Geoffroy P. Intranasal administration of crushed ALO-02 (extended-release oxycodone with sequestered naltrexone): A randomized, controlled abuse-potential study in nondependent recreational opioid users. J Clin Pharmacol. 2015 Dec;55(12):1351-61. doi: 10.1002/jcph.552. Epub 2015 Jul 2. PMID 26011742
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4531009&StudyName=A%20Study%20to%20Characterize%20the%20Abuse%20Liability%20of%20ALO-02%20in%20Healthy%2C%20Non-Dependent%2C%20Recreational%20Opioid%20Users%20When%20ALO-02%20Capsules%20are%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recreational opioid users who had experience with intranasal administration of opiates and were not dependent on opioids based on Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision (DSM-IV-TR) criteria, were recruited in this study.
Pre-assignment Details: After successful naloxone challenge test, all participants underwent training sessions involving complete pharmacodynamics test battery before the drug discrimination phase, to ensure that participants fully understood how to perform the tests, were comfortable, and attained a stable level of performance on the various performance-based measures.
Groups:
- Naloxone: Naloxone hydrochloride (HCl) 0.2 milligram (mg) intravenously followed by additional 0.6 mg naloxone hydrochloride intravenously on Day 0, each dose followed by an assessment for signs and symptoms of opioid withdrawal. Participants who did not display signs and symptoms of opioid withdrawal, were assigned to either oxycodone HCl 30 mg then placebo or placebo then oxycodone HCl 30 mg group in the drug discrimination phase of the study.
- Oxycodone HCl 30 mg Then Placebo: Single dose of oxycodone HCl 30 mg crushed tablet intranasally on Day 1 followed by single dose of placebo matched to oxycodone HCl 30 mg crushed tablet intranasally on Day 2. Participants were assigned to receive oxycodone HCl 30 mg and naltrexone HCl 3.6 mg extended-release (ALO-02) 30 mg/3.6 mg crushed capsule, placebo matched to ALO-02 30 mg/3.6 mg crushed capsule (placebo sugar spheres, PBO SS), oxycodone 30 mg crushed tablet (OXY 30 mg), placebo matched to oxycodone 30 mg crushed tablet (placebo lactose tablet, PBO Lac), intranasally, in any of the 4 sequences in the treatment phase of the study.
- Placebo Then Oxycodone HCl 30 mg: Single dose of placebo matched to oxycodone HCl 30 mg crushed tablet intranasally on Day 1 followed by single dose of oxycodone HCl 30 mg crushed tablet intranasally on Day 2. Participants were assigned to receive ALO-02 30 mg/3.6 mg crushed capsule, placebo matched to ALO-02 30 mg/3.6 mg crushed capsule (PBO SS), oxycodone 30 mg crushed tablet (OXY 30 mg), placebo matched to oxycodone 30 mg crushed tablet (PBO Lac), intranasally, in any of the 4 sequences in the treatment phase of the study.
- PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS: Single dose of placebo matched to oxycodone (PBO Lac) 30 mg crushed tablet intranasally in first intervention period; followed by single dose of oxycodone HCl 30 mg (OXY 30 mg) crushed tablet intranasally in second intervention period; then single dose of ALO-02 30 mg/3.6 mg crushed capsule intranasally in third intervention period; then single dose of placebo matched to ALO-02 (PBO SS) 30 mg/3.6 mg capsule intranasally in fourth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
- ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg: Single dose of ALO-02 30 mg/3.6 mg crushed capsule intranasally in first intervention period; followed by single dose of placebo matched to oxycodone (PBO Lac) 30 mg crushed tablet intranasally in second intervention period; then single dose of placebo matched to ALO-02 (PBO SS) 30 mg/3.6 mg crushed capsule intranasally in third intervention period; then single dose of oxycodone HCl 30 mg (OXY 30 mg) crushed tablet intranasally in fourth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
- OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg: Single dose of oxycodone HCl 30 mg (OXY 30 mg) crushed tablet intranasally in first intervention period; followed by single dose of placebo matched to ALO-02 (PBO SS) 30 mg/3.6 mg crushed capsule intranasally in second intervention period; then single dose of placebo matched to oxycodone (PBO Lac) 30 mg crushed tablet intranasally in third intervention period; then single dose of ALO-02 30 mg/3.6 mg crushed capsule intranasally in fourth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
- PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac: Single dose of placebo matched to ALO-02 (PBO SS) 30 mg/3.6 mg crushed capsule intranasally in first intervention period; followed by single dose of ALO-02 30 mg/3.6 mg crushed capsule intranasally in second intervention period; then single dose of oxycodone HCl 30 mg (OXY 30 mg) crushed tablet intranasally in third intervention period; then single dose of placebo matched to oxycodone (PBO Lac) 30 mg crushed tablet intranasally in fourth intervention period. A washout period of at least 5 days (not exceeding 14 days) was maintained between each intervention period.
Period: Naloxone Challenge Phase
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 45 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 45 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Drug Discrimination Phase: Day 1
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 0 | 22 | 23 | 0 | 0 | 0 | 0
Completed | 0 | 19 | 23 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 0 | 0 | 0 | 0
Period: Drug Discrimination Phase: Day 2
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 0 | 19 | 23 | 0 | 0 | 0 | 0
Completed | 0 | 16 | 16 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 7 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Did Not Meet Entrance Criteria | 0 | 2 | 7 | 0 | 0 | 0 | 0
Period: Treatment Phase: First Intervention
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 0 | 0 | 0 | 8 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Washout Period 1
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 0 | 0 | 0 | 8 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 8 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Phase: Second Intervention
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 0 | 0 | 0 | 8 | 8 | 7 | 8
Completed | 0 | 0 | 0 | 8 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Washout Period 2
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 0 | 0 | 0 | 8 | 8 | 7 | 8
Completed | 0 | 0 | 0 | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Phase: Third Intervention
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 0 | 0 | 0 | 7 | 8 | 7 | 8
Completed | 0 | 0 | 0 | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Washout Period 3
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 0 | 0 | 0 | 7 | 8 | 7 | 8
Completed | 0 | 0 | 0 | 6 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 1
Period: Treatment Phase: Fourth Intervention
Arm/Group | Naloxone | Oxycodone HCl 30 mg Then Placebo | Placebo Then Oxycodone HCl 30 mg | PBO Lac, OXY 30 mg, ALO-02 30 mg, PBO SS | ALO-02 30 mg, PBO Lac, PBO SS, OXY 30 mg | OXY 30 mg, PBO SS, PBO Lac, ALO-02 30 mg | PBO SS, ALO-02 30 mg, OXY 30 mg, PBO Lac
Started | 0 | 0 | 0 | 6 | 8 | 7 | 7
Completed | 0 | 0 | 0 | 6 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug, beginning with the naloxone challenge phase.
Groups:
- Entire Study Population: Included all participants enrolled in the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Drug Liking: Peak Effect (Emax)
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the extreme left with "strong disliking" (score of 0 mm) and on the extreme right with "strong liking" (score of 100 mm). Peak Effect (Emax) = Maximum observed score.
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: Completer analysis set included all randomized participants who completed all 4 periods of treatment phase and who contributed to post-dose Pharmacodynamic (PD) data from each period.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Placebo Sugar Spheres: Single dose of placebo matched to ALO-02 crushed capsule intranasally in any of the first to fourth intervention periods.
- ALO-02 30 mg: Single dose of ALO-02 30 mg/3.6 mg crushed capsule intranasally in any of the first to fourth intervention periods.
- Placebo Lactose Tablet: Single dose of placebo matched to oxycodone crushed tablet intranasally in any of the first to fourth intervention periods.
- Oxycodone 30 mg: Single dose of oxycodone HCl 30 mg crushed tablet intranasally in any of the first to fourth intervention periods.
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 50.9 (1.18) | 60.5 (12.05) | 51.3 (3.32) | 92.8 (11.98)
Statistical Analysis 1: Comparison: Placebo Sugar Spheres vs ALO-02 30 mg; Mixed-effect model with treatment, period, and sequence as fixed effects, and participants nested within the sequence as a random effect; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; Least Squares (LS) mean Difference = 9.5, 95% CI 2-sided [4.8 to 14.2]
Statistical Analysis 2: Comparison: ALO-02 30 mg vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = -32.3, 95% CI 2-sided [-37.0 to -27.6]
Statistical Analysis 3: Comparison: ALO-02 30 mg vs Placebo Lactose Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 9.1, 95% CI 2-sided [4.5 to 13.8]
Statistical Analysis 4: Comparison: Placebo Sugar Spheres vs Placebo Lactose Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8806, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = -0.4, 95% CI 2-sided [-5.0 to 4.3]
Statistical Analysis 5: Comparison: Placebo Lactose Tablet vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 41.4, 95% CI 2-sided [36.8 to 46.1]
Statistical Analysis 6: Comparison: Placebo Sugar Spheres vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 41.8, 95% CI 2-sided [37.1 to 46.4]

2. Primary Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-2 Hour
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the extreme left with "strong disliking" (score of 0 mm) and on the extreme right with "strong liking" (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hours.
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm | 98.518 (6.7606) | 105.286 (21.3736) | 100.241 (3.3227) | 159.580 (32.1643)
Statistical Analysis 1: Comparison: Placebo Sugar Spheres vs ALO-02 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2176, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 6.6, 95% CI 2-sided [-4.0 to 17.1]
Statistical Analysis 2: Comparison: ALO-02 30 mg vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = -54.6, 95% CI 2-sided [-65.1 to -44.1]
Statistical Analysis 3: Comparison: ALO-02 30 mg vs Placebo Lactose Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3502, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 5.0, 95% CI 2-sided [-5.6 to 15.5]
Statistical Analysis 4: Comparison: Placebo Sugar Spheres vs Placebo Lactose Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7624, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = -1.6, 95% CI 2-sided [-12.1 to 8.9]
Statistical Analysis 5: Comparison: Placebo Lactose Tablet vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 59.6, 95% CI 2-sided [49.0 to 70.1]
Statistical Analysis 6: Comparison: Placebo Sugar Spheres vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 61.2, 95% CI 2-sided [50.6 to 71.7]

3. Primary Outcome: High: Peak Effect (Emax)
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 2.2 (10.01) | 26.6 (28.44) | 6.0 (21.84) | 85.8 (24.34)
Statistical Analysis 1: Comparison: Placebo Sugar Spheres vs ALO-02 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 24.5, 95% CI 2-sided [13.8 to 35.3]
Statistical Analysis 2: Comparison: ALO-02 30 mg vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = -61.7, 95% CI 2-sided [-72.6 to -50.9]
Statistical Analysis 3: Comparison: ALO-02 30 mg vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 18.2, 95% CI 2-sided [7.4 to 29.1]
Statistical Analysis 4: Comparison: Placebo Sugar Spheres vs Placebo Lactose Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2507, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = -6.3, 95% CI 2-sided [-17.2 to 4.5]
Statistical Analysis 5: Comparison: Placebo Lactose Tablet vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 79.9, 95% CI 2-sided [69.2 to 90.7]
Statistical Analysis 6: Comparison: Placebo Sugar Spheres vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 86.3, 95% CI 2-sided [75.4 to 97.1]

4. Primary Outcome: High: Area Under Effect Curve (AUE) From 0-2 Hour
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hours.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm | 0.871 (3.5082) | 27.750 (39.7213) | 4.768 (20.0468) | 135.670 (43.0513)
Statistical Analysis 1: Comparison: Placebo Sugar Spheres vs ALO-02 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 26.9, 95% CI 2-sided [10.6 to 43.1]
Statistical Analysis 2: Comparison: ALO-02 30 mg vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = -109.3, 95% CI 2-sided [-125.7 to -93.0]
Statistical Analysis 3: Comparison: ALO-02 30 mg vs Placebo Lactose Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0109, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 21.4, 95% CI 2-sided [5.1 to 37.8]
Statistical Analysis 4: Comparison: Placebo Sugar Spheres vs Placebo Lactose Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5117, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = -5.4, 95% CI 2-sided [-21.8 to 10.9]
Statistical Analysis 5: Comparison: Placebo Lactose Tablet vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 130.8, 95% CI 2-sided [114.5 to 147.0]
Statistical Analysis 6: Comparison: Placebo Sugar Spheres vs Oxycodone 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was adjusted using Benjamini-Hochberg method; LS Mean Difference = 136.2, 95% CI 2-sided [119.8 to 152.5]

5. Secondary Outcome: Take Drug Again: Peak Effect (Emax)
Description: Take drug again VAS is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm VAS with score ranging from 0 mm to 100 mm (score of 0 mm = "definitely would not", 50 mm = "do not care", and 100 mm = "definitely would"). Emax = Maximum observed score.
Time Frame: Intervention period: 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 48.0 (14.91) | 58.3 (31.99) | 46.6 (18.75) | 87.8 (26.69)

6. Secondary Outcome: Take Drug Again: Mean Effect (Emean)
Description: Take drug again VAS is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm VAS with score ranging from 0 mm to 100 mm (score of 0 mm = "definitely would not", 50 mm = "do not care", and 100 mm = "definitely would"). Emean = Average observed score.
Time Frame: Intervention period: 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 44.71 (14.286) | 52.16 (30.926) | 43.95 (17.753) | 85.34 (26.860)

7. Secondary Outcome: Take Drug Again Effect at Hours 12 and 24
Description: Take drug again VAS is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm VAS with score ranging from 0 mm to 100 mm (score of 0 mm = "definitely would not", 50 mm = "do not care", and 100 mm = "definitely would").
Time Frame: Intervention period: 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm
  Hour 12 | 43.4 (17.36) | 51.5 (32.74) | 43.2 (18.02) | 87.4 (26.68)
  Hour 24 | 46.1 (17.40) | 52.8 (32.62) | 44.7 (20.66) | 83.3 (28.34)

8. Secondary Outcome: Overall Drug Liking: Peak Effect (Emax)
Description: Overall drug liking VAS assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carry-over effects). A 100 mm VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm = "neither like nor dislike", and 100 mm= "strong liking"). Emax = Maximum observed score.
Time Frame: Intervention period: 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 50.5 (0.84) | 59.9 (21.70) | 51.5 (6.59) | 85.1 (23.84)

9. Secondary Outcome: Overall Drug Liking: Mean Effect (Emean)
Description: Overall drug liking VAS assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carry-over effects). A 100 mm VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm = "neither like nor dislike", and 100 mm= "strong liking"). Emean = Average observed score.
Time Frame: Intervention period: 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 50.32 (0.641) | 56.77 (20.058) | 49.16 (8.131) | 81.25 (24.081)

10. Secondary Outcome: Overall Drug Liking Effect at Hours 12 and 24
Description: Overall drug liking VAS assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carry-over effects). A 100 mm VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm = "neither like nor dislike", and 100 mm= "strong liking").
Time Frame: Intervention period: 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm
  Hour 12 | 50.3 (0.53) | 56.0 (20.69) | 50.5 (2.28) | 81.8 (25.73)
  Hour 24 | 50.4 (0.87) | 57.6 (21.34) | 47.8 (15.02) | 80.8 (25.05)

11. Secondary Outcome: Any Drug Effects: Peak Effect (Emax)
Description: Any Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 0.6 (1.42) | 35.5 (31.81) | 6.2 (17.51) | 88.6 (21.28)

12. Secondary Outcome: Any Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour and 0-24 Hour
Description: Any Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm
  AUE (0-1) | 0.295 (1.0179) | 18.647 (21.1164) | 1.692 (7.6048) | 69.692 (21.7465)
  AUE (0-2) | 0.429 (1.5517) | 38.290 (43.2746) | 3.701 (16.0503) | 138.888 (48.0836)
  AUE (0-8) | 0.830 (2.4083) | 82.371 (117.8336) | 12.513 (54.8407) | 329.004 (197.0154)
  AUE (0-24) | 1.045 (2.5917) | 96.013 (138.6860) | 12.585 (54.8265) | 399.719 (311.1514)

13. Secondary Outcome: Any Drug Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Any Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours | 0.267 [0.25 to 24.02] | 0.517 [0.25 to 12.02] | 0.250 [0.23 to 8.00] | 0.267 [0.25 to 3.02]

14. Secondary Outcome: Good Drug Effects: Peak Effect (Emax)
Description: Good Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 4.3 (13.70) | 25.6 (29.60) | 8.4 (17.98) | 87.9 (21.04)

15. Secondary Outcome: Good Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour and 0-24 Hour
Description: Good Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm
  AUE (0-1) | 0.804 (3.3233) | 14.263 (20.5630) | 2.393 (9.4972) | 69.464 (21.0703)
  AUE (0-2) | 0.902 (3.5146) | 26.603 (39.6360) | 5.161 (20.4142) | 138.679 (45.7222)
  AUE (0-8) | 2.777 (10.0925) | 58.746 (110.6803) | 14.795 (62.5301) | 307.589 (191.3034)
  AUE (0-24) | 6.420 (28.9445) | 69.246 (136.6847) | 14.795 (62.5301) | 348.732 (274.1036)

16. Secondary Outcome: Good Drug Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Good Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours | 0.267 [0.25 to 8.02] | 0.275 [0.25 to 2.52] | 0.250 [0.23 to 3.00] | 0.400 [0.25 to 1.52]

17. Secondary Outcome: Bad Drug Effects: Peak Effect (Emax)
Description: Bad Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 1.4 (5.49) | 13.0 (24.52) | 5.6 (15.92) | 18.5 (26.24)

18. Secondary Outcome: Bad Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour and 0-24 Hour
Description: Bad Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm
  AUE (0-1) | 0.045 (0.1674) | 3.911 (7.8416) | 0.246 (1.2050) | 4.080 (9.9234)
  AUE (0-2) | 0.116 (0.4053) | 6.920 (12.0601) | 0.701 (3.6120) | 10.107 (21.5289)
  AUE (0-8) | 0.482 (1.5766) | 15.000 (31.8735) | 5.719 (20.3316) | 43.232 (87.5335)
  AUE (0-24) | 6.696 (32.9731) | 19.214 (45.0219) | 6.004 (20.3044) | 71.375 (192.3920)

19. Secondary Outcome: Bad Drug Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Bad Drug Effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours | 0.267 [0.25 to 24.02] | 0.267 [0.25 to 2.52] | 0.250 [0.23 to 12.00] | 0.642 [0.25 to 12.02]

20. Secondary Outcome: Feel Sick: Peak Effect (Emax)
Description: Feel Sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: Intervention periods: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 2.1 (9.23) | 8.7 (20.50) | 3.9 (13.34) | 4.6 (21.95)

21. Secondary Outcome: Feel Sick: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour and 0-24 Hour
Description: Feel Sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm
  AUE (0-1) | 0.036 (0.1438) | 1.549 (5.3704) | 0.232 (1.2041) | 0.442 (1.5106)
  AUE (0-2) | 0.545 (2.3162) | 3.424 (8.1912) | 0.714 (3.6100) | 3.049 (8.5600)
  AUE (0-8) | 1.170 (4.6220) | 9.371 (22.4283) | 4.804 (19.8483) | 25.103 (80.5454)
  AUE (0-24) | 1.313 (4.6839) | 10.513 (24.8145) | 4.875 (19.8377) | 42.460 (144.3171)

22. Secondary Outcome: Feel Sick: Time to Maximum (Peak) Effect (TEmax)
Description: Feel Sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours | 0.267 [0.25 to 4.00] | 0.267 [0.25 to 6.00] | 0.250 [0.23 to 8.00] | 0.267 [0.25 to 8.02]

23. Secondary Outcome: Nausea: Peak Effect (Emax)
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 1.9 (9.25) | 9.3 (20.99) | 5.3 (15.90) | 12.3 (29.94)

24. Secondary Outcome: Nausea: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour and 0-24 Hour
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm
  AUE (0-1) | 0.036 (0.1477) | 2.455 (5.9882) | 0.290 (1.2186) | 2.339 (6.0186)
  AUE (0-2) | 0.473 (2.3127) | 5.179 (11.0690) | 0.781 (3.6209) | 7.357 (15.8889)
  AUE (0-8) | 1.000 (4.6313) | 9.063 (17.1052) | 5.353 (19.5238) | 46.402 (114.6615)
  AUE (0-24) | 1.071 (4.6706) | 10.848 (23.1275) | 5.638 (19.5807) | 58.759 (150.9858)

25. Secondary Outcome: Nausea: Time to Maximum (Peak) Effect (TEmax)
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours | 0.267 [0.25 to 4.02] | 0.267 [0.25 to 6.00] | 0.250 [0.23 to 2.52] | 0.267 [0.25 to 8.02]

26. Secondary Outcome: Sleepy: Peak Effect (Emax)
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 7.6 (21.35) | 35.0 (36.04) | 11.1 (28.41) | 62.9 (36.25)

27. Secondary Outcome: Sleepy: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour and 0-24 Hour
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm
  AUE (0-1) | 0.813 (2.6613) | 8.848 (13.8043) | 2.920 (6.8778) | 20.464 (21.9449)
  AUE (0-2) | 2.580 (7.9968) | 34.571 (40.4452) | 8.089 (19.0222) | 61.750 (48.0978)
  AUE (0-8) | 19.518 (52.5582) | 125.196 (157.0183) | 34.438 (92.1369) | 304.652 (210.8188)
  AUE (0-24) | 26.875 (60.2903) | 187.839 (217.5872) | 64.795 (172.8842) | 496.652 (424.7570)

28. Secondary Outcome: Sleepy: Time to Maximum (Peak) Effect (TEmax)
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours | 0.267 [0.25 to 12.02] | 1.517 [0.25 to 12.02] | 0.267 [0.25 to 12.02] | 2.517 [0.25 to 12.02]

29. Secondary Outcome: Dizzy: Peak Effect (Emax)
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
mm | 4.4 (13.34) | 7.4 (15.74) | 4.1 (15.02) | 23.5 (36.62)

30. Secondary Outcome: Dizzy: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour and 0-24 Hour
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm
  AUE (0-1) | 0.036 (0.1890) | 1.161 (2.7284) | 0.795 (3.1320) | 9.192 (14.5426)
  AUE (0-2) | 0.482 (2.3628) | 5.134 (14.4253) | 1.259 (4.6194) | 17.737 (28.2806)
  AUE (0-8) | 3.286 (10.6279) | 8.482 (20.2822) | 4.938 (22.2685) | 48.826 (93.0141)
  AUE (0-24) | 7.143 (28.6404) | 11.768 (29.2486) | 5.152 (22.2481) | 57.469 (119.5335)

31. Secondary Outcome: Dizzy: Time to Maximum (Peak) Effect (TEmax)
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours | 0.267 [0.25 to 8.02] | 0.267 [0.25 to 12.02] | 0.250 [0.23 to 24.02] | 0.267 [0.25 to 6.00]

32. Secondary Outcome: Percentage of Dose (Drug Powder) Insufflated
Description: The percentage of dose insufflated, was based on a calculation of the weight of powder remaining (if any) following each dosing during the intervention period.
Time Frame: Intervention period: 0 Hour post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 29 | 30 | 30 | 32
percentage of dose | 100.00 (0.000) | 99.85 (0.840) | 100.00 (0.000) | 99.37 (3.553)

33. Secondary Outcome: Pupillometry: Peak Effect (Emax)
Description: Pupillometry assessments measure change in pupil size (miosis) as an indicator of opioid pharmacological properties. Participants have the size of pupil measured using a pupillometer. Measurements are made in a dimly lit (mesopic) room with controlled lighting conditions. The same eye for each participant was used for all measurements during the study. Emax = Maximum observed score.
Time Frame: Intervention period: pre-dose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: Completer analysis set included all randomized participants who completed all 4 periods of treatment phase and who contributed to post-dose PD data from each period. Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 26 | 28 | 26
mm | -0.9 (0.60) | -1.7 (0.64) | -0.7 (0.50) | -2.9 (0.66)

34. Secondary Outcome: Pupillometry: Area Under Effect Curve (AUE) From 0-1 Hour, 0-2 Hour, 0-8 Hour and 0-24 Hour
Description: Pupillometry assessments measure change in pupil size (miosis) as an indicator of opioid pharmacological properties. Participants have the size of pupil measured using a pupillometer. Measurements are made in a dimly lit (mesopic) room with controlled lighting conditions. The same eye for each participant was used for all measurements during the study. AUE (0-x) = Area under the effect versus time curve from time zero to time of last quantifiable effect (0-x).
Time Frame: Intervention period: pre-dose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: Completer analysis set included all randomized participants who completed all 4 periods of treatment phase and who contributed to post-dose Pharmacodynamic (PD) data from each period. Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 26 | 28 | 26
hours*mm
  AUE (0-1) | 5.333 (0.8204) | 4.746 (0.8291) | 5.132 (0.7712) | 3.229 (0.4547)
  AUE (0-2) | 10.538 (1.7478) | 9.114 (1.6974) | 10.162 (1.5217) | 5.868 (0.8325)
  AUE (0-8) | 42.623 (6.9054) | 34.874 (6.6910) | 41.658 (6.0399) | 23.904 (3.3208)
  AUE (0-24) | 130.666 (18.7096) | 110.574 (19.3751) | 128.937 (16.8685) | 94.012 (12.6818)

35. Secondary Outcome: Pupillometry: Time to Maximum (Peak) Effect (TEmax)
Description: Pupillometry assessments measure change in pupil size (miosis) as an indicator of opioid pharmacological properties. Participants have the size of pupil measured using a pupillometer. Measurements are made in a dimly lit (mesopic) room with controlled lighting conditions. The same eye for each participant was used for all measurements during the study. TEmax = Time to maximum observed score.
Time Frame: Intervention period: pre-dose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 34
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 26 | 28 | 26
hours | 3.017 [0.53 to 24.03] | 3.017 [0.53 to 12.02] | 2.025 [0.53 to 24.03] | 0.800 [0.52 to 3.03]

36. Other Pre Specified Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-1 Hour, 0-8 Hour and 0-24 Hour
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time 0 to x hours (0-x).
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm
  AUE (0-1) | 49.143 (4.2752) | 53.455 (10.0825) | 49.884 (2.7778) | 81.250 (13.1291)
  AUE (0-8) | 395.455 (17.5470) | 414.045 (61.6430) | 401.036 (3.4801) | 540.554 (122.5684)
  AUE (0-24) | 1198.955 (18.4210) | 1223.902 (72.4917) | 1202.750 (6.0623) | 1397.911 (231.2330)

37. Other Pre Specified Outcome: Drug Liking: Time to Maximum (Peak) Effect (TEmax)
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Intervention period: 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours | 0.383 [0.25 to 3.02] | 0.758 [0.25 to 8.00] | 0.500 [0.23 to 6.02] | 0.383 [0.25 to 12.02]

38. Other Pre Specified Outcome: High: Area Under Effect Curve (AUE) From 0-1 Hour, 0-8 Hour and 0-24 Hours
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-x) = Area under the effect versus time curve from time 0 to x hours (0-x).
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours*mm
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours*mm
  AUE (0-1) | 0.790 (3.3474) | 14.250 (20.4883) | 2.313 (9.3978) | 68.223 (19.7926)
  AUE (0-8) | 1.049 (3.8560) | 60.143 (113.5249) | 12.955 (51.4525) | 290.670 (174.8869)
  AUE (0-24) | 1.121 (4.0488) | 75.429 (136.4319) | 16.598 (70.5151) | 330.813 (257.7739)

39. Other Pre Specified Outcome: High: Time to Maximum (Peak) Effect (TEmax)
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 28 | 28 | 28 | 28
hours | 0.258 [0.25 to 0.52] | 0.275 [0.25 to 24.00] | 0.250 [0.23 to 3.00] | 0.517 [0.25 to 2.03]

40. Other Pre Specified Outcome: Subject Rating Scale for Nasal Effects: Peak Effect (Emax)
Description: Participant-rated scale for nasal effects was used to assess burning, need to blow nose, runny nose/nasal discharge, facial pain/pressure, and nasal congestion using a 6-point scale (where, 0 = not present/no problem; 1 = very mild problem; 2 = mild/slight problem; 3 = moderate problem; 4 = severe problem; 5 = problem "as bad as can be"). Emax = Maximum observed score.
Time Frame: Intervention period: pre-dose, 0.5, 0.75, 1, 1.5, 2 hours post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 29 | 30 | 30 | 32
units on a scale
  Burning | 0.0 (0.00) | 0.1 (0.25) | 0.0 (0.32) | 0.5 (0.88)
  Need to Blow Nose | 0.1 (0.37) | 0.1 (0.61) | 0.1 (0.51) | 0.4 (0.80)
  Runny Nose/ Nasal Discharge | 0.0 (0.33) | 0.1 (0.57) | 0.3 (0.98) | 0.4 (0.84)
  Facial Pain/ Pressure | 0.0 (0.19) | 0.0 (0.26) | 0.1 (0.37) | 0.3 (0.67)
  Nasal Congestion | 0.1 (0.46) | 0.2 (0.77) | 0.4 (1.10) | 0.4 (0.84)

41. Other Pre Specified Outcome: Subject Rating Scale for Nasal Effects: Area Under Effect Curve (AUE) From 0-1 Hour and 0-2 Hour
Description: Participant-rated scale for nasal effects was used to assess burning, need to blow nose, runny nose/nasal discharge, facial pain/pressure, and nasal congestion using a 6-point scale (where, 0 = not present/no problem; 1 = very mild problem; 2 = mild/slight problem; 3 = moderate problem; 4 = severe problem; 5 = problem "as bad as can be"). AUE (0-x) = Area under the effect versus time curve from time 0 to x hours (0-x).
Time Frame: Intervention period: pre-dose, 0.5, 0.75, 1, 1.5, 2 hours post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale*hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 29 | 30 | 30 | 32
units on a scale*hours
  Burning: AUE (0-1) | 0.000 (0.0000) | 0.025 (0.0951) | 0.033 (0.1035) | 0.184 (0.3062)
  Burning: AUE (0-2) | 0.000 (0.0000) | 0.025 (0.0951) | 0.033 (0.1035) | 0.270 (0.6214)
  Need to Blow Nose: AUE (0-1) | 0.129 (0.3125) | 0.117 (0.3182) | 0.088 (0.2503) | 0.293 (0.4586)
  Need to Blow Nose: AUE (0-2) | 0.164 (0.4147) | 0.183 (0.5520) | 0.088 (0.2503) | 0.504 (0.8616)
  Runny Nose/ Nasal Discharge: AUE (0-1) | 0.069 (0.2468) | 0.083 (0.3432) | 0.038 (0.1046) | 0.184 (0.3521)
  Runny Nose/ Nasal Discharge: AUE (0-2) | 0.086 (0.3342) | 0.108 (0.4437) | 0.146 (0.4678) | 0.301 (0.6771)
  Facial Pain/ Pressure: AUE (0-1) | 0.009 (0.0464) | 0.033 (0.1428) | 0.042 (0.1367) | 0.066 (0.2057)
  Facial Pain/ Pressure: AUE (0-2) | 0.009 (0.0464) | 0.050 (0.2312) | 0.050 (0.1416) | 0.184 (0.6270)
  Nasal Congestion: AUE (0-1) | 0.172 (0.4111) | 0.175 (0.3664) | 0.200 (0.3934) | 0.250 (0.3269)
  Nasal Congestion: AUE (0-2) | 0.259 (0.6399) | 0.250 (0.5835) | 0.242 (0.4956) | 0.484 (0.7853)

42. Other Pre Specified Outcome: Subject Rating Scale for Nasal Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Participant-rated scale for nasal effects was used to assess burning, need to blow nose, runny nose/nasal discharge, facial pain/pressure, and nasal congestion using a 6-point scale (where, 0 = not present/no problem; 1 = very mild problem; 2 = mild/slight problem; 3 = moderate problem; 4 = severe problem; 5 = problem "as bad as can be"). TEmax = Time to maximum observed score.
Time Frame: Intervention period: pre-dose, 0.5, 0.75, 1, 1.5, 2 hours post-dose
Population: as for baseline characteristics
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 29 | 30 | 30 | 32
hours
  Burning | 0.517 [0.50 to 0.53] | 0.517 [0.50 to 0.60] | 0.517 [0.48 to 0.55] | 0.517 [0.50 to 1.52]
  Need to Blow Nose | 0.517 [0.50 to 0.53] | 0.517 [0.50 to 0.60] | 0.517 [0.48 to 0.55] | 0.517 [0.50 to 1.52]
  Runny Nose/ Nasal Discharge | 0.517 [0.50 to 0.53] | 0.517 [0.50 to 0.75] | 0.517 [0.48 to 1.52] | 0.517 [0.50 to 1.52]
  Facial Pain/ Pressure | 0.517 [0.50 to 0.53] | 0.517 [0.50 to 0.60] | 0.517 [0.48 to 2.00] | 0.517 [0.50 to 1.52]
  Nasal Congestion | 0.517 [0.50 to 0.53] | 0.517 [0.50 to 0.75] | 0.517 [0.48 to 0.78] | 0.525 [0.50 to 1.52]

43. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax) of Oxycodone, Oxymorphone and Noroxycodone
Description: Participants who received oxycodone and ALO-02 were reported. Oxymorphone and noroxycodone are metabolites of oxycodone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: Parameter analysis set included all enrolled participants who received at least 1 dose of study drug and who had at least 1 of the pharmacokinetic (PK) parameters of interest.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | ALO-02 30 mg | Oxycodone 30 mg
Number analyzed (Participants) | 30 | 32
nanogram per milliliter (ng/mL)
  Oxycodone | 57.93 (13.706) | 82.63 (19.877)
  Oxymorphone | 0.4613 (0.25684) | 0.3441 (0.16644)
  Noroxycodone | 29.02 (10.858) | 18.88 (6.8506)

44. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax) of Naltrexone and 6-beta-naltrexol
Description: Participants who received ALO-02 were reported. 6-Beta-naltrexol is metabolites of naltrexone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: Parameter analysis set included all enrolled participants who received at least 1 dose of study drug and who had at least 1 of the PK parameters of interest.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | ALO-02 30 mg
Number analyzed (Participants) | 30
nanogram per milliliter (ng/mL)
  Naltrexone | 4.574 (1.4093)
  6-beta-naltrexol | 4.085 (1.2948)

45. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Oxycodone, Oxymorphone and Noroxycodone
Description: Participants who received oxycodone and ALO-02 were reported. Oxymorphone and noroxycodone are metabolites of oxycodone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: Parameter analysis set included all enrolled participants who received at least 1 dose of study drug and who had at least 1 of the PK parameters of interest. Here 'n' signifies participants evaluable for specified category for each arm, respectively.
Measure: Median (Full Range); unit: hours
Arm/Group | ALO-02 30 mg | Oxycodone 30 mg
Number analyzed (Participants) | 30 | 32
hours
  Oxycodone (n = 30, 32) | 1.59 [0.283 to 4.07] | 0.475 [0.283 to 1.07]
  Oxymorphone (n = 29, 32) | 2.05 [1.05 to 4.07] | 2.55 [0.550 to 6.03]
  Noroxycodone (n = 30, 32) | 2.08 [1.05 to 6.08] | 4.05 [2.05 to 6.10]

46. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Naltrexone and 6-beta-naltrexol
Description: Participants who received ALO-02 were reported. 6-Beta-naltrexol is metabolites of naltrexone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 44
Measure: Median (Full Range); unit: hours
Arm/Group | ALO-02 30 mg
Number analyzed (Participants) | 30
hours
  Naltrexone | 0.317 [0.283 to 1.57]
  6-Beta-naltrexol | 2.05 [0.767 to 4.07]

47. Other Pre Specified Outcome: Plasma Decay Half-Life (t1/2) of Oxycodone, Oxymorphone and Noroxycodone
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Participants who received oxycodone and ALO-02 were reported. Oxymorphone and noroxycodone are metabolites of oxycodone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ALO-02 30 mg | Oxycodone 30 mg
Number analyzed (Participants) | 30 | 32
hours
  Oxycodone (n = 30, 32) | 4.171 (0.65437) | 4.134 (0.87884)
  Oxymorphone (n = 1, 1) | NA (NA) — Data was not reported when fewer than 3 participant were evaluable. | NA (NA) — Data was not reported when fewer than 3 participant were evaluable.
  Noroxycodone (n = 28, 27) | 7.116 (1.2582) | 7.101 (0.89387)

48. Other Pre Specified Outcome: Plasma Decay Half-Life (t1/2) of Naltrexone and 6-beta-naltrexol
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Participants who received ALO-02 were reported. 6-Beta-naltrexol is metabolites of naltrexone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: Parameter analysis set included all enrolled participants who received at least 1 dose of study drug and who had at least 1 of the PK parameters of interest. Here 'n' signifies those participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ALO-02 30 mg
Number analyzed (Participants) | 30
hours
  Naltrexone (n = 30) | 3.577 (0.71124)
  6-beta-naltrexol (n = 11) | 9.230 (0.62809)

49. Other Pre Specified Outcome: Area Under the Concentration-Time Curve (AUC) From 0-1 Hour, 0-2 Hour and 0-8 Hour of Oxycodone, Oxymorphone and Noroxycodone
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. Participants who received oxycodone and ALO-02 were reported. Oxymorphone and noroxycodone are metabolites of oxycodone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8 hours post-dose
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | ALO-02 30 mg | Oxycodone 30 mg
Number analyzed (Participants) | 30 | 32
nanogram*hour/milliliter (ng*hr/mL)
  Oxycodone: AUC (0-1) | 33.59 (10.010) | 59.56 (14.977)
  Oxycodone: AUC (0-2) | 81.26 (21.951) | 116.3 (27.449)
  Oxycodone: AUC (0-8) | 263.9 (64.753) | 328.2 (73.834)
  Oxymorphone: AUC (0-1) | 0.09544 (0.07603) | 0.1589 (0.10643)
  Oxymorphone: AUC (0-2) | 0.4023 (0.26464) | 0.4211 (0.25186)
  Oxymorphone: AUC (0-8) | 1.979 (1.1448) | 1.856 (0.99704)
  Noroxycodone: AUC (0-1) | 5.726 (4.0397) | 6.410 (2.8655)
  Noroxycodone: AUC (0-2) | 26.37 (15.014) | 18.91 (7.1716)
  Noroxycodone: AUC (0-8) | 147.7 (46.804) | 119.9 (40.380)

50. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Oxycodone, Oxymorphone and Noroxycodone
Description: Area under the plasma concentration time-curve from zero to the last quantifiable concentration (AUClast). Participants who received oxycodone and ALO-02 were reported. Oxymorphone and noroxycodone are metabolites of oxycodone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | ALO-02 30 mg | Oxycodone 30 mg
Number analyzed (Participants) | 30 | 32
nanogram*hour/milliliter (ng*hr/mL)
  Oxycodone | 353.0 (103.13) | 435.3 (112.11)
  Oxymorphone | 2.498 (1.6933) | 2.469 (1.8058)
  Noroxycodone | 280.6 (95.277) | 248.5 (84.723)

51. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Oxycodone, Oxymorphone and Noroxycodone
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). Participants who received oxycodone and ALO-02 were reported. Oxymorphone and noroxycodone are metabolites of oxycodone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | ALO-02 30 mg | Oxycodone 30 mg
Number analyzed (Participants) | 30 | 32
nanogram*hour/milliliter (ng*hr/mL)
  Oxycodone (n = 30, 32) | 361.2 (109.33) | 447.3 (123.92)
  Oxymorphone (n = 1, 1) | NA (NA) — Data was not reported when fewer than 3 participant were evaluable. | NA (NA) — Data was not reported when fewer than 3 participant were evaluable.
  Noroxycodone (n = 28, 27) | 309.9 (111.42) | 288.8 (104.33)

52. Other Pre Specified Outcome: Area Under the Concentration-Time Curve (AUC) From 0-1 Hour, 0-2 Hour and 0-8 Hour of Naltrexone and 6-beta-naltrexol
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. Participants who received ALO-02 were reported. 6-Beta-naltrexol is metabolites of naltrexone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8 hours post-dose
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | ALO-02 30 mg
Number analyzed (Participants) | 30
nanogram*hour/milliliter (ng*hr/mL)
  Naltrexone: AUC (0-1) | 3.127 (0.87457)
  Naltrexone: AUC (0-2) | 5.669 (1.4721)
  Naltrexone: AUC (0-8) | 10.25 (3.0400)
  6-beta-naltrexol: AUC (0-1) | 1.050 (0.56296)
  6-beta-naltrexol: AUC (0-2) | 3.862 (1.7302)
  6-beta-naltrexol: AUC (0-8) | 18.78 (4.8024)

53. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Naltrexone and 6-beta-naltrexol
Description: Area under the plasma concentration time-curve from zero to the last quantifiable concentration (AUClast). Participants who received ALO-02 were reported. 6-Beta-naltrexol is metabolites of naltrexone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | ALO-02 30 mg
Number analyzed (Participants) | 30
nanogram*hour/milliliter (ng*hr/mL)
  Naltrexone | 11.07 (3.2130)
  6-beta-naltrexol | 37.28 (9.3207)

54. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Naltrexone and 6-beta-naltrexol
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). Participants who received ALO-02 were reported. 6-Beta-naltrexol is metabolites of naltrexone.
Time Frame: Intervention period: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | ALO-02 30 mg
Number analyzed (Participants) | 30
nanogram*hour/milliliter (ng*hr/mL)
  Naltrexone (n = 11) | 10.71 (11.13)
  6-beta-naltrexol (n = 30) | 45.85 (10.544)

55. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 3 - 7 days following last study drug administration that were absent before treatment or that worsened relative to pre-treatment state. Symptoms of withdrawal following naloxone administration (naloxone challenge phase) were not collected as adverse events unless they met the criteria for an SAE. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Screening up to 3 to 7 days following last study drug administration, or time of early withdrawal
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Naloxone: Naloxone HCl 0.2 mg intravenously followed by additional 0.6 mg naloxone HCl intravenously, each dose followed by an assessment for signs and symptoms of opioid withdrawal in naloxone challenge phase.
- Oxycodone HCl 30 mg: Single dose of oxycodone HCl 30 mg crushed tablet intranasally on either of 2 days in drug discrimination phase.
- Placebo Oxycodone HCl: Single dose of placebo matched to oxycodone HCl 30 mg crushed tablet intranasally on either of 2 days in drug discrimination phase.
- Placebo Sugar Spheres: Single dose of placebo matched to ALO-02 30 mg/3.6 mg crushed capsule intranasally in any of the first to fourth intervention periods.
- Placebo Lactose Tablet: Single dose of placebo matched to oxycodone 30 mg crushed tablet intranasally in any of the first to fourth intervention periods.
Arm/Group | Naloxone | Oxycodone HCl 30 mg | Placebo Oxycodone HCl | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 45 | 45 | 42 | 29 | 30 | 30 | 32
participants
  AEs | 1 | 43 | 8 | 6 | 18 | 10 | 32
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

56. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change in Vital Sign Examinations
Description: Vital signs assessment included measurement of heart rate, systolic and diastolic blood pressures, and respiratory rate. Criteria for clinically significant change in any vital sign examination was based on investigator's discretion.
Time Frame: Screening up to 3 to 7 days following last study drug administration, or time of early withdrawal
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Naloxone | Oxycodone HCl 30 mg | Placebo Oxycodone HCl | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 45 | 45 | 42 | 29 | 30 | 30 | 32
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

57. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change in End Tidal Carbon Dioxide (EtCO2)
Description: End-tidal carbon dioxide concentration in the expired air (EtCO2) was monitored using capnography in a sitting position. Criteria for clinically significant change in EtCO2 was based on investigator's discretion.
Time Frame: Intervention period: pre-dose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 29 | 30 | 30 | 32
participants | 0 | 0 | 0 | 0

58. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change in Oxygen Saturation of Hemoglobin (SpO2)
Description: Oxygen saturation of hemoglobin in blood (SpO2) was monitored using pulse oximetry continuously for 5 hours following dosing in the drug discrimination phase and continuously for 12 hours following dosing in the treatment phase, or longer at the discretion of the investigator. Individual measurement was collected in a sitting position. If SpO2 fall below 90 percent (%), the investigator administered oxygen via nasal cannula at a flow rate sufficient to maintain the SpO2 greater than or equal to 90%. Participants with fall in SpO2 below 90% were reported.
Time Frame: Drug discrimination phase: pre-dose up to 5 hours; intervention period: pre-dose up to 12 hours
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Oxycodone HCl 30 mg | Placebo Oxycodone HCl | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Number analyzed (Participants) | 45 | 42 | 29 | 30 | 30 | 32
participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Naloxone | Oxycodone HCl 30 mg | Placebo Oxycodone HCl | Placebo Sugar Spheres | ALO-02 30 mg | Placebo Lactose Tablet | Oxycodone 30 mg
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/42 | 0/29 | 0/30 | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 1/45 | 43/45 | 3/45 | 4/29 | 16/30 | 7/30 | 32/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naloxone (N=45) | Oxycodone HCl 30 mg (N=45) | Placebo Oxycodone HCl (N=45) | Placebo Sugar Spheres (N=29) | ALO-02 30 mg (N=30) | Placebo Lactose Tablet (N=30) | Oxycodone 30 mg (N=32)
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 6 | 0 | 0 | 2 | 0 | 5
Fatigue (General disorders) | 0 | 8 | 0 | 1 | 4 | 2 | 3
Feeling hot (General disorders) | 0 | 6 | 0 | 0 | 2 | 0 | 3
Feeling of relaxation (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 7 | 1 | 0 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 6 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 3 | 3 | 3
Somnolence (Nervous system disorders) | 0 | 20 | 1 | 1 | 4 | 1 | 12
Euphoric mood (Psychiatric disorders) | 0 | 41 | 2 | 1 | 10 | 0 | 27
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 24 | 1 | 0 | 0 | 0 | 24
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.